CLINICAL TRIAL: NCT04611997
Title: Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With Lymph Node Dissection for Locally Advanced Gastric Cancer After Neoadjuvant Chemotherapy
Brief Title: IGG Using in Laparoscopic Gastrectomy for Locally Advanced Gastric Cancer After Neoadjuvant Chemotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-020
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Gastric Cancer; Lymph Node Metastases
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Group A (Study Group): Laparoscopic gastrectomy group with the use of near-infrared imaging (ICG group) Group B (Control Group): Laparoscopic gastrectomy group without the use of near-infrared imaging (Non-ICG group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Laparoscopic gastrectomy group with the use of near-infrared imaging (ICG group)
  Interventions: Drug: Indocyanine Green
- Group B (Placebo Comparator): Laparoscopic gastrectomy group without the use of near-infrared imaging (Non-ICG group)
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — Indocyanine Green Tracer Using in Laparoscopic Gastrectomy with Lymph Node Dissection for Locally Advanced Gastric Cancer After Neoadjuvant

SUMMARY:
Patients with locally advanced gastric adenocarcinoma (cT2-4a N-/+ M0) were selected as study subjects to investigate the safety, efficacy, and feasibility of ICG near-infrared imaging tracing in guiding laparoscopic D2 lymph node dissection for gastric cancer after neoadjuvant chemotherapy by comparing injection ICG group and non-injection ICG group

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT2-4a, N-/+, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual, 8th Edition
4. No distant metastasis, no invasion of pancreas, spleen or other adjacent organs in the preoperative examinations
5. Performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) score I to III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous gastric surgery (including ESD/EMR for gastric cancer)
5. Enlarged or bulky regional lymph node (diameter over 3cm) supported by preoperative imaging.
6. Other malignant disease within the past 5 years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within past six months
9. History of cerebrovascular accident within past six months
10. History of continuous systematic administration of corticosteroids within one month
11. Requirement for simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1 (forced expiratory volume in one second)<50% of predicted values
14. Diffuse invasive gastric cancer
15. Preoperatively, tumors involving the squamocolumnar junction or duodenum were confirmed
16. A history of iodine allergy
17. Refuse laparoscopic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 3 years
  Disease-free survival is calculated from the day of surgery to the day of recurrence (When the specific date of recurrence of the tumor is unknown, the ending point is the date of death due to tumor causes). In the event that neither death nor recurrence of the tumor are observed, the end point is the final date that a patient is confirmed as relapse-free.

SECONDARY OUTCOMES:
Total number of retrieved lymph nodes | 30 days
  Total number of retrieved lymph nodes

CONTACTS AND LOCATIONS:
Locations (1):
- Chang-ming Huang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided